CLINICAL TRIAL: NCT00231049
Title: A Phase 1 Trial Evaluating Safety, Tolerability and Immune Response of AG-707 Compared to Placebo in HSV-2 Seropositive Patients
Brief Title: Trial Evaluating Safety, Tolerability and Immune Response of AG-707
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Agenus Inc. (Industry)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: C-400-01
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Last update posted 2008-10-27 (Estimated); Status verified 2008-10

CONDITIONS: Genital Herpes
Keywords: Genital Herpes; HSV-2 Seropositive; Vaccine
MeSH Terms: conditions — Herpes Genitalis

INTERVENTIONS:
Drug: AG-707

SUMMARY:
This is a randomized, multi-center, sequential, dose-escalating study of three dose cohorts of AG-707. Individuals who meet all of the inclusion and exclusion criteria for eligibility will be randomized to receive either AG-707 (at the 80 µg dose), AG-707 with QS-21 (at the 80 µg dose), placebo, or QS-21. Each patient will be monitored for safety as specified in the protocol.

DETAILED DESCRIPTION:
Primary Objective:

Determine the overall safety profile of three different dose levels of AG-707 vaccination (with and without an adjuvant, QS-21) at 80, 240 and 400 µg compared to placebo and QS-21 alone in HSV-2 seropositive adults.

Secondary Objective:

Determine immune response to AG-707 vaccination (with and without QS-21) at dose cohorts of 80, 240, and 400 µg as compared to placebo and QS-21 alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be seropositive for HSV-2 (+/- HSV-1) and have a documented history of clinically active genital herpes (at least one prior outbreak).
* Patients must be seronegative for HIV.
* Patients must be seronegative for hepatitis B and C
* Have baseline chemistry and hematology (hemoglobin, white blood cell (WBC), absolute neutrophil count (ANC), eosinophils) within normal limits; prothrombin time (PT) and partial thromboplastin time (PTT) below the upper limit of normal (ULN), and platelets above the lower limit of normal (LLN). Basophils, lymphocytes and monocytes must be within 1.2 x ULN or 0.8 x LLN and considered not clinically significant by the investigator. Total creatine phosphokinase (CPK) laboratory values < 1.25X the upper limit of normal (according to the normal reference ranges of the Central Laboratory) at baseline (Screening and Pre-Study Visit) and considered not clinically significant by the Investigator.
* Patients must not be taking antiviral therapy.
* Must be between the ages of 18 and 50 years of age and willing to either use an effective method of contraception or abstain from sexual activity for the 28-week duration of the trial.

Exclusion Criteria:

* Severe active infection, compromised cardiopulmonary function, or other serious medical illness that, in the opinion of the Principal Investigator, would prevent study completion.
* History of HSV infection of the eye (herpes simplex interstitial keratitis or uveitis), or herpes-associated erythema multiforme.
* History of immune suppression or autoimmune disorder.
* Concomitant use of systemic corticosteroids or other immunosuppressive medications (including nasal and inhaled steroids). The use of nasal steroids for seasonal rhinitis is acceptable.
* Patients with known hypersensitivity or allergies to acyclovir or valacyclovir.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2006-03

PRIMARY OUTCOMES:
Determine the overall safety profile of three different dose levels of AG-707 vaccination (with and without an adjuvant, QS-21) at 80, 240 and 400 µg compared to placebo and QS-21 alone in herpes simplex virus-2 (HSV-2) seropositive adults

SECONDARY OUTCOMES:
Determine immune response to AG-707 vaccination (with and without QS-21) at dose cohorts of 80, 240, and 400 µg as compared to placebo and QS-21 alone

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Indianapolis, Indiana
  - Portland, Oregon
  - Seattle, Washington